CLINICAL TRIAL: NCT00210158
Title: Effects of Intraoperative Nitrous Oxide on Postoperative Pain for Patients With Current Opioid Treatment After Vertebroplasty.
Brief Title: Intraoperative Nitrous Oxide and Postoperative Pain for Patients With Current Opioid Treatment
Acronym: PROTOX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IB2005-05
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Chronic Pain
Keywords: Current opioid treatment; Nitrous oxide; Chronic pain; Opioid therapy; Postoperative hyperalgesia; Acute opioid tolerance
MeSH Terms: conditions — Chronic Pain | interventions — Air; Protoporphyrinogen Oxidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air arm (Reference) (Sham Comparator): Patients undergo long-term morphine treatment and vertebral cementoplasty. During the procedure, patients are ventilated with a mixture of air and oxygen.
  Interventions: Procedure: Air
- Protox Arm (Experimental) (Experimental): Patients undergo long-term morphine treatment and vertebral cementoplasty. During the procedure, patients are ventilated with a mixture of oxygen and nitrous oxide.
  Interventions: Procedure: Protox

INTERVENTIONS:
Procedure: Air — Patients undergo long-term morphine treatment and vertebral cementoplasty. During the procedure, patients are ventilated with a mixture of air and oxygen.
  Arms: Air arm (Reference)
Procedure: Protox — Patients undergo long-term morphine treatment and vertebral cementoplasty. During the procedure, patients are ventilated with a mixture of oxygen and nitrous oxide.
  Arms: Protox Arm (Experimental)

SUMMARY:
Peroperative opioids are known to induce N-Methyl-D-Aspartate dependent enhancement of postoperative hyperalgesia. For patients with current opioid treatment, these phenomena could be exagerated and could produce greater postoperative opioid consumption and higher pain score. Since Nitrous oxide has anti- N-Methyl-D-Aspartate properties, the aim of this study was to evaluate, in patients with current opioid treatment, the effects of peroperative Nitous oxide on postoperative opioid consumption and pain score, after vertebroplasty.

ELIGIBILITY:
* Older than 18 years
* Current opioid treatment > 1 month
* patients scheduled to undergo vertebroplasty with general anesthesia

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2006-12-31 (Actual); Study Completion 2006-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Lakdja, MD, Principal Investigator — Institut Bergonié
Locations (1):
- Institut Bergonié - Centre Régional de Luttre Contre le Cancer DE Bordeaux et du Sud Ouest, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Air Arm (Reference) | Protox Arm (Experimental)
Started | 19 | 20
Completed | 19 | 18
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Air Arm (Reference) | Protox Arm (Experimental) | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (2.8) | 63.6 (2.7) | 62.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Post-operative Morphine Consumption
Description: Morphine consumption (mg) during PCA (Patient Controlled Analgesia)
Time Frame: Between surgery and up to 48 hours
Population: Participants with a record of morphine consumption (mg) during PCA (Patient Controlled Analgesia)
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Air Arm (Reference) | Protox Arm (Experimental)
Number analyzed (Participants) | 18 | 18
mg | 54.6 (51.2) | 44.8 (46.4)
Statistical Analysis 1: Comparison: Air Arm (Reference) vs Protox Arm (Experimental); T-test for a difference of means, assuming independant samples and unequal variances; Test type: Superiority; p = 0.5, t-test, 2 sided; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [-23.4 to 42.8]

2. Secondary Outcome: Proportion of Participants With Post-operative Pain
Description: Pain is measured using a visual analog scale (VAS), ranging from 0 (no pain) to 100 (worst pain ever).
  A participant is considered to have pain if VAS score is >= 40.
Time Frame: Between surgery and up to 48 hours
Population: Participants with a VAS score record available.
Measure: Count of Participants; unit: Participants
Arm/Group | Air Arm (Reference) | Protox Arm (Experimental)
Number analyzed (Participants) | 19 | 16
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: 48 hours
Arm/Group | Air Arm (Reference) | Protox Arm (Experimental)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 0/19 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes